CLINICAL TRIAL: NCT02712996
Title: Treatment Outcomes With Lisdexamfetamine Dimesylate (Vyvanse) in Children With Traumatic Brain Injury-Related Attention Deficits
Brief Title: Treatment of Traumatic Brain Injury (TBI)-Related Attention Deficits in Children
Acronym: TBIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Michael G. Tramontana, Ph.D., Associate Professor of Psychiatry and Neurology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TBI 56592
Record Dates: First submitted 2016-03-08; First posted 2016-03-18 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Traumatic Brain Injury; Attention Deficit Disorder
Keywords: Traumatic Brain Injury; Attention Deficit; TBI; Vyvanse
MeSH Terms: conditions — Brain Injuries, Traumatic; Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vyvanse (Active Comparator): Lisdexamfetamine (Vyvanse) capsule, 20-70 mg, each morning for 6 weeks.
  Interventions: Drug: Lisdexamfetamine
- Placebo (Placebo Comparator): Placebo capsule, 20-70 mg, each morning for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine — Lisdexamfetamine (Vyvanse) capsule, 20-70 mg, each morning for 6 weeks.
  Other Names: Vyvanse
  Arms: Vyvanse
Drug: Placebo — Placebo capsule, 20-70 mg, each morning for 6 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this research study is to evaluate whether Vyvanse, a psychostimulant, can help children ages 6-16 with attention deficits due to traumatic brain injury (TBI). Vyvanse is currently approved for the treatment of Attention-Deficit/Hyperactivity (ADHD). The exact effects this drug may have on adults with attention deficits caused by TBI have been investigated prior. The exact effects this drug may have on children with attention deficits caused by TBI are not known, but the investigators expect that Vyvanse will be of some help in treating this population as well.

DETAILED DESCRIPTION:
Symptoms of inattentiveness, impulsivity, and poor persistence have been observed in children following traumatic brain injury (TBI). These often are among the most prominent symptoms manifested and may contribute to interference in a variety of other functional domains. Although there has been some use of psychostimulant medication to treat TBI-acquired attention deficits, it remains a relatively uncommon clinical practice. This study, by highlighting mechanisms of action, could serve to promote the appropriate use of this type of treatment for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 6 to 16
* Traumatic brain injury rated as mild/moderate/severe (based on Glasgow Coma Scale, estimated posttraumatic amnesia, indications of intracranial injury on CT scan, etc.)
* Sustained 2-36 months earlier
* Considered to be neurologically stable (absence of post-acute symptoms of confusion, disorientation, etc.)
* Persistent (> 2 months) problems with focused or sustained attention
* Problems with attention/concentration rated as among the most prominent cognitive changes
* Accompanying features may include diminished arousal/speed/stamina and/or hyperactivity/impulsivity symptoms.

Exclusion Criteria:

* Cases with primarily penetrating head trauma
* Pre-injury history of diagnosed ADHD
* Pre-injury history of other neurodevelopmental disorders including intellectual disabilities, major communication disorders, autism spectrum disorder
* Unstable or serious psychiatric conditions, such as psychotic symptoms. Concurrent problems with depression, anxiety, or post-traumatic stress disorder may be present but are judged to be stable and not so severe as to require pharmacologic treatment
* Treatment with psychotropic medication(s), including psychostimulant(s) within the last 6 months, but eligible thereafter
* Lifetime history of stimulant abuse or dependence. Other (non-stimulant) substance abuse within the past 6 months.
* Tics or other contraindications for psychostimulant use including cardiovascular disease, uncontrolled hypertension or hyperthyroidism, glaucoma, agitation, use of an monoamine oxidase (MAO) inhibitor within the past six weeks. Pregnancy would also be an exclusion for girls of childbearing age.
* Estimated intelligence quotient (IQ) < 70
* Sensory and/or motor impairment(s) seriously limiting testing options
* Neurological conditions including uncontrolled epilepsy, degenerative disorders, brain tumor, or stroke
* Physical condition affecting arousal, activity level, or stamina including uncontrolled thyroid dysfunction, severe or symptomatic anemia, autoimmune or metabolic disorders, untreated moderate/severe sleep apnea, etc.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Tramontana, Ph.D, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 20 enrolled participants, 3 never began the trial due to scheduling problems or competing demands.
Groups:
- Lisdexamfetamine (Vyvanse) Then Placebo: Participants first received Lisdexamfetamine (Vyvanse) capsule, 20-70 mg, each morning for 6 weeks. On day 43 after treatment initiation, each subject was switched to placebo capsule, 20-70 mg, each morning for 6 weeks.
- Placebo Then Vyvanse: Participants first received Placebo capsule, 20-70 mg, each morning for 6 weeks. On day 43 after treatment initiation, participants received Lisdexamfetamine (Vyvanse) capsule, 20-70 mg, each morning for 6 weeks
Period: First Intervention (Study Days 1-42)
Arm/Group | Lisdexamfetamine (Vyvanse) Then Placebo | Placebo Then Vyvanse
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: Second Intervention (Study Days 43-84)
Arm/Group | Lisdexamfetamine (Vyvanse) Then Placebo | Placebo Then Vyvanse
Started | 8 | 9
Completed | 8 | 8
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lisdexamfetamine (Vyvanse) Then Placebo: Participants first received Lisdexamfetamine (Vyvanse) capsule, 20-70 mg, each morning for 6 weeks. Then on day 43 after treatment initiation, each subject received Placebo capsule, 20-70 mg, each morning for 6 weeks
- Placebo Then Lisdexamfetamine (Vyvanse): Participants first received Placebo capsule, 20-70 mg, each morning for 6 weeks. Then on day 43 after treatment initiation, each subject received Lisdexamfetamine (Vyvanse) capsule, 20-70 mg, each morning for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Lisdexamfetamine (Vyvanse) Then Placebo | Placebo Then Lisdexamfetamine (Vyvanse) | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 9 | 17
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessing Severity of Symptoms Associated With Attention-deficit/Hyperactivity Disorder (ADHD) in Children When Using Vyvanse Versus Placebo by Administering the Conners-3 Parent Form
Description: The Conners-3 Parent Form is used to obtain the parent's observations about behavior in their child aged 6 to 18 years old. Parents rate the child's behavior on 45 items as not true at all (0) to very much true (3). The lowest scale score is 0 (better behavior) and the highest is 135 (worse behavior). The Conners 3-P includes content Scales of Inattention, Hyperactivity/Impulsivity, Learning Problems, Executive Functioning, Aggression, and Peer/Family Relations. Inattention scale was reported as the Primary Outcome. All scores were converted to z-scores (M=0, SD=+/-1).
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Lisdexamfetamine (Vyvanse): Participants who received Lisdexamfetamine (Vyvanse) capsule, 20-70 mg, each morning in either the or last 6 weeks of the study.
- Placebo: Participants who received Placebo capsule, 20-70 mg, each morning in either the or last 6 weeks of the study.
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 1.00 (1.11) | 1.76 (1.47)

2. Primary Outcome: Assessing Executive Functioning in Children When Using Vyvanse Versus Placebo by Administering the Behavior Rating Inventory of Executive Function (BRIEF) - PARENT
Description: The BRIEF Parent Questionnaire is a validated 86-item questionnaire composed of 8 clinical scales that measure different aspects of executive functioning (Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor, Inhibit, Shift, Emotional Control). For each item, parents rate whether the child engages in the behavior "never" (=1), "sometimes" (=2), or "often" (=3). The lowest scale score is 86 (better performance) and the highest is 258 (worse performance). The clinical scales form two broader Indexes (Behavioral Regulation and Metacognition) and an overall score, the Global Executive Composite (GEC). GEC was reported as the Primary Outcome. Raw scores were converted to z-scores (M=0, SD=+/-1).
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.51 (0.99) | 1.16 (1.33)

3. Primary Outcome: Assessing Inattentiveness in Children Using Vyvanse Versus Placebo by Measuring Omissions on the Conners Continuous Performance Task (CPT-II).
Description: Conner's Continuous Performance Task (CPT-II) measures sustained attention and response inhibition. During the CPT-II, letters were presented serially on a screen in a random order. All letters were considered target stimuli, except for the letter 'X' which is a non-target stimulus. Participants responded to target stimuli by pressing the space bar of a computer keyboard (90% of the stimuli) while withholding responses to non-target stimuli (10% of the test). Omission errors represented the number of times a participant fails to respond to target letters (all other than 'X'). Raw scores were converted to z-scores (M=0, SD=+/-1). Higher scores indicate greater inattentiveness.
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 16 | 17
Z score | 0.63 (1.71) | 1.33 (1.68)

4. Primary Outcome: Assessing Physical Symptoms in Children Using Vyvanse Versus Placebo by Measuring Anxiety on the Revised Child Manifest Anxiety Scale (RCMAS)
Description: RCMAS is a self-report, 37-item questionnaire in which children agree (yes = 1) or disagree (no =0) to statements about themselves. A Total Anxiety score is computed based on 28 items, which are divided into 3 anxiety subscales: physiological anxiety (10 items), worry/oversensitivity (11 items), and social concerns/concentration (7 items). The remaining nine items on the RCMAS constitute the Lie (social desirability) subscale. The lowest scale score is 0 and the highest is 37. Raw scores were converted to z-scores (M=0, SD=+/-1). Because scores are derived from affirmative responses, a high score indicates a high level of anxiety or lie on that subscale.
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.12 (0.79) | -0.23 (0.95)

5. Primary Outcome: Assessing Total Symptoms in Children Using Vyvanse Versus Placebo by Measuring Anxiety on the Revised Child Manifest Anxiety Scale (RCMAS)
Description: as for outcome 4
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | -0.3 (0.85) | -0.56 (0.89)

6. Primary Outcome: Assessing Attention Problems in Children Using Vyvanse Versus Placebo by Measuring Symptoms on the Child Behavior Checklist (CBCL)
Description: The Child Behavior Checklist (CBCL) is a widely used caregiver report form identifying problem behavior in children. The patient is rated on 113 items scored on a 3-point Likert scale (0=not true; 1=somewhat/sometimes true; 2=very true/often true). CBCL consists of eight empirically-based syndrome subscales. The range of subscale scores (summed) are: Aggressive Behavior (0-36), Anxious/Depressed (0-26), Attention Problems (0-20), Rule-Breaking Behavior (0-34), Somatic Complaints (0-22), Social Problems (0-22), Thought Problems (0-30), and Withdrawn/Depressed (0-16). Raw scores were converted to z-scores (M=0, SD=+/-1). Higher scores indicate more severe symptoms.
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.88 (0.69) | 1.37 (0.93)

7. Primary Outcome: Assessing Anxiety-Depression Problems in Children Using Vyvanse Versus Placebo by Measuring Symptoms on the Child Behavior Checklist (CBCL)
Description: as for outcome 6
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.44 (0.52) | 0.76 (0.66)

8. Primary Outcome: Assessing Inhibitory Control in Children When Using Vyvanse Versus Placebo Utilizing the Inhibit Subscale on the Behavior Rating Inventory of Executive Function (BRIEF) - PARENTS
Description: The BRIEF Parent Questionnaire is a validated 86-item questionnaire composed of 8 clinical scales that measure different aspects of executive functioning (Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor, Inhibit, Shift, Emotional Control). For each item, parents rate whether the child engages in the behavior "never" (=1), "sometimes" (=2), or "often" (=3). The lowest scale score is 86 (better performance) and the highest is 258 (worse performance). The clinical scales form two broader Indexes (Behavioral Regulation and Metacognition) and an overall score, the Global Executive Composite (GEC). Inhibit was reported as the Primary Outcome. Raw scores were converted to z-scores (M=0, SD=+/-1).
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | -0.05 (1.05) | 0.42 (1.16)

9. Primary Outcome: Assessing Ability to Tolerate Change in Children When Using Vyvanse Versus Placebo by Utilizing the Shift Subscale on the Behavior Rating Inventory of Executive Function (BRIEF) - PARENTS
Description: The BRIEF Parent Questionnaire is a validated 86-item questionnaire composed of 8 clinical scales that measure different aspects of executive functioning (Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor, Inhibit, Shift, Emotional Control). For each item, parents rate whether the child engages in the behavior "never" (=1), "sometimes" (=2), or "often" (=3). The lowest scale score is 86 (better performance) and the highest is 258 (worse performance). The clinical scales form two broader Indexes (Behavioral Regulation and Metacognition) and an overall score, the Global Executive Composite (GEC). Shift was reported as the Primary Outcome. Raw scores were converted to z-scores (M=0, SD=+/-1).
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.33 (1.22) | 1 (1.44)

10. Primary Outcome: Assessing Ability to Begin Tasks in Children When Using Vyvanse Versus Placebo by Utilizing the Initiate Subscale on the Behavior Rating Inventory of Executive Function (BRIEF) - PARENTS
Description: The BRIEF Parent Questionnaire is a validated 86-item questionnaire composed of 8 clinical scales that measure different aspects of executive functioning (Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor, Inhibit, Shift, Emotional Control). For each item, parents rate whether the child engages in the behavior "never" (=1), "sometimes" (=2), or "often" (=3). The lowest scale score is 86 (better performance) and the highest is 258 (worse performance). The clinical scales form two broader Indexes (Behavioral Regulation and Metacognition) and an overall score, the Global Executive Composite (GEC). Initiate was reported as the Primary Outcome. Raw scores were converted to z-scores (M=0, SD=+/-1).
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.64 (0.89) | 1.23 (1.04)

11. Primary Outcome: Assessing Representational Memory in Children When Using Vyvanse Versus Placebo by Utilizing the Working Memory Subscale on the Behavior Rating Inventory of Executive Function (BRIEF) - PARENTS
Description: The BRIEF Parent Questionnaire is a validated 86-item questionnaire composed of 8 clinical scales that measure different aspects of executive functioning (Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor, Inhibit, Shift, Emotional Control). For each item, parents rate whether the child engages in the behavior "never" (=1), "sometimes" (=2), or "often" (=3). The lowest scale score is 86 (better performance) and the highest is 258 (worse performance). The clinical scales form two broader Indexes (Behavioral Regulation and Metacognition) and an overall score, the Global Executive Composite (GEC). Working Memory was reported as the Primary Outcome. Raw scores were converted to z-scores (M=0, SD=+/-1).
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.96 (1.25) | 1.69 (1.26)

12. Primary Outcome: Assessing Task-oriented Monitoring in Children When Using Vyvanse Versus Placebo by Utilizing the Monitor Subscale on the Behavior Rating Inventory of Executive Function (BRIEF) - PARENTS
Description: The BRIEF Parent Questionnaire is a validated 86-item questionnaire composed of 8 clinical scales that measure different aspects of executive functioning (Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor, Inhibit, Shift, Emotional Control). For each item, parents rate whether the child engages in the behavior "never" (=1), "sometimes" (=2), or "often" (=3). The lowest scale score is 86 (better performance) and the highest is 258 (worse performance). The clinical scales form two broader Indexes (Behavioral Regulation and Metacognition) and an overall score, the Global Executive Composite (GEC). Monitor was reported as the Primary Outcome. Raw scores were converted to z-scores (M=0, SD=+/-1).
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.34 (0.89) | 0.84 (1.19)

13. Primary Outcome: Assessing Behavior Regulation in Children When Using Vyvanse Versus Placebo by Measuring the Behavior Regulation Index (BRI) on the Behavior Rating Inventory of Executive Function (BRIEF) - PARENTS
Description: The BRIEF Parent Questionnaire is a validated 86-item questionnaire composed of 8 clinical scales that measure different aspects of executive functioning (Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor, Inhibit, Shift, Emotional Control). For each item, parents rate whether the child engages in the behavior "never" (=1), "sometimes" (=2), or "often" (=3). The lowest scale score is 86 (better performance) and the highest is 258 (worse performance). The clinical scales form two broader Indexes (Behavioral Regulation and Metacognition) and an overall score, the Global Executive Composite (GEC). Behavior Regulation was reported as the Primary Outcome. Raw scores were converted to z-scores (M=0, SD=+/-1).
Time Frame: 12 weeks
Population: All participants who received at least one dose of each intervention were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | -0.04 (1.12) | 0.48 (1.21)

14. Primary Outcome: Assessing Cognitive Regulation in Children When Using Vyvanse Versus Placebo by Measuring the Cognitive Regulation Index (CRI) on the Behavior Rating Inventory of Executive Function (BRIEF) - PARENTS
Description: The BRIEF Parent Questionnaire is a validated 86-item questionnaire composed of 8 clinical scales that measure different aspects of executive functioning (Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor, Inhibit, Shift, Emotional Control). For each item, parents rate whether the child engages in the behavior "never" (=1), "sometimes" (=2), or "often" (=3). The lowest scale score is 86 (better performance) and the highest is 258 (worse performance). The clinical scales form two broader Indexes (Behavioral Regulation and Metacognition) and an overall score, the Global Executive Composite (GEC). Cognitive Regulation was reported as the Primary Outcome. Raw scores were converted to z-scores (M=0, SD=+/-1).
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.68 (1.02) | 1.33 (1.31)

15. Primary Outcome: Assessing Emotion Regulation in Children When Using Vyvanse Versus Placebo by Measuring the Emotion Regulation Index (ERI) on the Behavior Rating Inventory of Executive Function (BRIEF) - PARENTS
Description: The BRIEF Parent Questionnaire is a validated 86-item questionnaire composed of 8 clinical scales that measure different aspects of executive functioning (Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor, Inhibit, Shift, Emotional Control). For each item, parents rate whether the child engages in the behavior "never" (=1), "sometimes" (=2), or "often" (=3). The lowest scale score is 86 (better performance) and the highest is 258 (worse performance). The clinical scales form two broader Indexes (Behavioral Regulation and Metacognition) and an overall score, the Global Executive Composite (GEC). Emotion regulation was reported as the Primary Outcome. Raw scores were converted to z-scores (M=0, SD=+/-1).
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.35 (1.16) | 0.94 (1.39)

16. Primary Outcome: Assessing Hyperactivity in Children When Using Vyvanse Versus Placebo by Administering the Conners-3 Parent Form
Description: The Conners-3 Parent Form is used to obtain the parent's observations about behavior in their child aged 6 to 18 years old. Parents rate the child's behavior on 45 items as not true at all (0) to very much true (3). The lowest scale score is 0 (better behavior) and the highest is 135 (worse behavior). The Conners 3-P includes content Scales of Inattention, Hyperactivity/Impulsivity, Learning Problems, Executive Functioning, Aggression, and Peer/Family Relations. Hyperactivity was reported as the Primary Outcome. All scores were converted to z-scores (M=0, SD=+/-1).
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.075 (1.45) | 0.71 (1.56)

17. Primary Outcome: Assessing Executive Functioning in Children When Using Vyvanse Versus Placebo by Administering the Conners-3 Parent Form
Description: The Conners-3 Parent Form is used to obtain the parent's observations about behavior in their child aged 6 to 18 years old. Parents rate the child's behavior on 45 items as not true at all (0) to very much true (3). The lowest scale score is 0 (better behavior) and the highest is 135 (worse behavior). The Conners 3-P includes content Scales of Inattention, Hyperactivity/Impulsivity, Learning Problems, Executive Functioning, Aggression, and Peer/Family Relations. Executive Functioning was reported as the Primary Outcome. All scores were converted to z-scores (M=0, SD=+/-1).Higher T-scores
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.97 (1.24) | 1.79 (1.58)

18. Secondary Outcome: Assessing Executive Functioning in Children When Using Vyvanse Versus Placebo by Administering the Behavior Rating Inventory of Executive Function (BRIEF) - CHILD SELF REPORT
Description: The BRIEF Self-Report Version assesses an adolescent's (ages 11-18) view of his or her cognitive, emotional, and behavioral functions. It is a validated 55-item questionnaire composed of 8 clinical scales that measure different aspects of executive functioning (Inhibit, Shift, Emotional Control, Monitor, Working Memory, Plan/Organize, Organization of Materials, and Task Completion). For each item, the child rates whether they engage in the behavior "never" (=1), "sometimes" (=2), or "often" (=3). The lowest scale score is 55 (better performance) and the highest is 165 (worse performance). The clinical scales form two broader Indexes (Behavioral Regulation and Metacognition) and an overall score, the Global Executive Composite (GEC). GEC was reported as the Primary Outcome. Raw scores were converted to z-scores (M=0, SD=+/-1).
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.66 (1.08) | 0.59 (1.14)

19. Secondary Outcome: Assessing Working Memory and Concentration in Children Using Vyvanse Versus Placebo by Measuring Performance on the Digit Span Subtest of the Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V)
Description: Digit Span repeats strings of digits of increasing length said by the examiner. Participants were asked to repeat the digits in the same sequence, either forwards or backwards. Every item on Digit Span consists of two trials. One point was awarded if the participant passed only 1 trial of a sequence length. Zero points were given if the participant failed both trials. It measures working memory and concentration with a range of scaled scores from 0-19. Raw scores were converted to z-scores (M=0, SD=+/-1). Higher scores indicate better recall and attention.
Time Frame: 12 weeks
Population: 1 participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | -0.27 (0.84) | -0.29 (1.01)

20. Secondary Outcome: Assessing Sustained Attention and Response Inhibition in Children Using Vyvanse Versus Placebo by Measuring Reaction Time (RT) Standard Error (SE) on the Conners Continuous Performance Task (CPT-II).
Description: Conner's Continuous Performance Task (CPT-II) measure sustained attention and response inhibition. During the CPT-II, letters were presented serially on a screen in a random order. All letters were considered target stimuli, except for the letter 'X' which is a non-target stimulus. Participants responded to target stimuli by pressing the space bar of a computer keyboard (90% of the stimuli) while withholding responses to non-target stimuli (10% of the test). Raw scores were converted to z-scores (M=0, SD=+/-1). Hit Reaction Time (RT) Standard Error (SE) measures response speed consistency. The higher the Overall Standard Error, the greater the inconsistency in the response speed, indicating a greater amount of inattention.
Time Frame: 12 weeks
Population: Missing data from 2 participants in the Placebo arm and 2 participants in the Vyvanse arm
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 14 | 15
Z-score | 0.14 (1.28) | 0.57 (1.53)

21. Secondary Outcome: Assessing Sustained Attention and Response Inhibition in Children Using Vyvanse Versus Placebo by Measuring RT Inter-Stimulus Interval (ISI) on the Conners Continuous Performance Task (CPT-II).
Description: Conner's Continuous Performance Task (CPT-II) measure sustained attention and response inhibition. During the CPT-II, letters were presented serially on a screen in a random order. All letters were considered target stimuli, except for the letter 'X' which is a non-target stimulus. Participants responded to target stimuli by pressing the space bar of a computer keyboard (90% of the stimuli) while withholding responses to non-target stimuli (10% of the test). CPT-II Hit Reaction Time (RT) Inter-Stimulus Interval (ISI) Change assesses the ability to adapt to changing inter-stimulus intervals. Inter-stimulus intervals refers to the amount of time between presentation of stimuli. High t-scores indicate that RT increased as the ISI increased; negative values indicate that RT decreased as the ISI increased.
  Less Hit RT ISI Change indicates less variability in RT depending on the speed of presentation.
Time Frame: 12 weeks
Population: This assessment was not administered.
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Assessing Sustained Attention and Response Inhibition in Children Using Vyvanse Versus Placebo by Measuring Hit Reaction Time (RT) Block Change on the Conners Continuous Performance Task (CPT-II).
Description: Conner's Continuous Performance Task (CPT-II) measures sustained attention and response inhibition. During the CPT-II, letters were presented serially on a screen in a random order. All letters were considered target stimuli, except for the letter 'X' which is a non-target stimulus. Participants responded to target stimuli by pressing the space bar of a computer keyboard (90% of the stimuli) while withholding responses to non-target stimuli (10% of the test). Raw scores were converted to z-scores (M=0, SD=+/-1). Overall hit reaction time is the average speed of correct responses for the entire test. Lower values indicate that responses got quicker as the test progressed. High values indicate a substantial slowing in reaction times.
Time Frame: 12 weeks
Population: 1 participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Vyvanse | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 0.75 (1.49) | 1.19 (1.39)

23. Secondary Outcome: Assessing Sustained Attention and Response Inhibition in Children Using Vyvanse Versus Placebo by Measuring Perseverations on the Conners Continuous Performance Task (CPT-II).
Description: Conner's Continuous Performance Task (CPT-II) measures sustained attention and response inhibition. During the CPT-II, letters were presented serially on a screen in a random order. All letters were considered target stimuli, except for the letter 'X' which is a non-target stimulus. Participants responded to target stimuli by pressing the space bar of a computer keyboard (90% of the stimuli) while withholding responses to non-target stimuli (10% of the test). CPT-II Perseverations represent responses in which reaction time was less than 100 ms; these responses are assumed to be anticipatory, random, or slow/inattentive (i.e., carried over from the previous response) because it is physiologically impossible to respond accurately in so short a time. Raw scores were converted to z-scores (M=0, SD=+/-1) to have them on a uniform metric. Higher scores indicate greater inattentiveness.
Time Frame: 12 weeks
Population: One participant completed the placebo arm, but dropped out of Vyvanse arm due to adverse event
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
Number analyzed (Participants) | 16 | 17
Z-score | 1.02 (1.89) | 0.86 (1.69)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Lisdexamfetamine (Vyvanse): Participants who received Lisdexamfetamine (Vyvanse) capsule, 20-70 mg, each morning in either the first or last 6 weeks of the study.
- Placebo: Participants who received Placebo capsule, 20-70 mg, each morning in either the first or last 6 weeks of the study.
Arm/Group | Lisdexamfetamine (Vyvanse) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 1/17 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine (Vyvanse) (N=17) | Placebo (N=17)
Anxiety (General disorders) | 1 (1) | 0 (0) — Increased anxiety, including panic-like symptoms,

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT02712996/Prot_SAP_000.pdf